CLINICAL TRIAL: NCT02369978
Title: Cardiovascular Health Investigation and Collaboration From Countries of America to Assess the Markers and Outcomes of Chagas Disease (CHICAMOCHA-3) - EQUITY (Equivalence of Usual Interventions for Trypanosomiasis)
Brief Title: CHICAMOCHA 3 - Equivalence of Usual Interventions for Trypanosomiasis (EQUITY)
Acronym: CHICAMOCHA-3
Status: Unknown | Phase: Phase 2 / Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Universidad Autónoma de Bucaramanga (Other)
Collaborators: Fundación Cardioinfantil Instituto de Cardiología (Other); Instituto Nacional de Salud, Colombia (Other Government); Instituto Nacional de Parasitologia Dr. Mario Fatala Chaben (Other Government)
Responsible Party: Principal Investigator, Juan Carlos Villar, MD, PhD, Professor, Department of Medicine, Universidad Autónoma de Bucaramanga
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 124156935014
Record Dates: First submitted 2015-02-17; First posted 2015-02-24 (Estimated); Last update posted 2017-07-21 (Actual); Status verified 2017-07

CONDITIONS: Chagas Disease
Keywords: Trypanocidal therapy; Benznidazole; Nifurtimox; Polymerase chain reaction; Randomized trial
MeSH Terms: conditions — Chagas Disease | interventions — Nifurtimox; benzonidazole; Control Groups

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Nifurtimox (NFX) (Experimental): 60 days of active treatment with full-dose, or 120 days of active treatment with half-dose (allocation ratio 1:1). The 60-day group will receive active treatment in the first or second half of a 120-day treatment window, as per random allocation. The active treatment period will be followed/preceded by matching placebo (see placebo arm below)
  Interventions: Drug: Nifurtimox
- Benznidazole (BZN) (Active Comparator): 60 days of active treatment with full-dose, or 120 days of active treatment with half-dose (allocation ratio 1:1). The 60-day group will receive active treatment in the first or second half of a 120-day treatment window, as per random allocation. The active treatment period will be followed/preceded by matching placebo (see placebo arm below)
  Interventions: Drug: Benznidazole
- Placebo (Placebo Comparator): 120 days of treatment with matching placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Nifurtimox — Full dose: 8 mg/Kg/day, assuming an average weight of 60 Kg: 240 mg B.I.D Half-dose: 120 mg B.I.D
  Other Names: Lampit (Bayer)
  Arms: Nifurtimox (NFX)
Drug: Benznidazole — Full dose: 5 mg/Kg/day, assuming an average weight of 60 Kg: 150 mg B.I.D Half dose: 75 mg B.I.D
  Other Names: Radanil (Roche), Rochagan (Roche), Abarax (ELEA)
  Arms: Benznidazole (BZN)
Drug: Placebo — Two capsules of matching placebo (contaning Magnesium stearate and cellulose) B.I.D
  Other Names: Control group
  Arms: Placebo

SUMMARY:
This randomized, blind, parallel-group trial will evaluate the efficacy and safety of Nifurtimox (NFX) and Benznidazole (BZN), the two usual interventions to treat the parasite Trypanosoma cruzi.

The investigators will test whether NFX is an effective trypanocidal agent (by comparison with placebo) and equivalent to BZN (as active comparator) in terms of both parasite-related and safety outcomes.

Individuals found seropositive and without clinical signs of dilated cardiomyopathy will receive either of the active treatments or matching placebo. Participants allocated to NFX or BZN will receive either a 60-day (full-dose) or a 120-day (half-dose) active treatment, whereas the control group will receive placebo for 120 days. There will be thus four arms of active treatment (NFX60, NFX120, BZN60 and BZN120), and a fifth control arm receiving placebo (1:1:1:1:1 allocation ratio) where every participant in the trial will take 120 days of study drug (the groups receiving full-dose will complete a 120-day masked treatment with placebo).

The study plans to enroll 500 participants from Colombia (in two different geographical areas) and Argentina, in order to explore regional differences in the treatment effects.

DETAILED DESCRIPTION:
The specific aims of this multi-center randomized trial include:

1. To evaluate the feasibility of conducting a multinational trial in terms of

   1. the ability to identify and recruit T. cruzi-infected individuals without clinical disease in a relatively short period
   2. the standardization of procedures to test the parasitic load using polymerase chain reaction (PCR)
2. To evaluate, in the study population, the efficacy of a treatment with NFX using conventional (full) dose (8/mg/Kg/day) or half-dose for a variable duration (full-dose for 60 days versus half-dose for 120 days) in terms of the presence of positive PCR tests one year after treatment, as compared with placebo.
3. To evaluate the equivalence (in terms of non-inferiority of its impact over the PCR testing) of two treatment schedules with NFX: a full-dose treatment for 60 days and a half-dose treatment for 120 days.
4. To evaluate the equivalence of two treatment schedules with BZN: A conventional (full) dose of 5 mg/Kg/day) for 60 days, as compared with half-dose treatment for 120 days.
5. To evaluate the equivalence of the treatment schedules with NFX as compared with those with BZN 5
6. To evaluate the safety (in terms of reporting of mild symptoms, limitation of daily activities or hospitalizations, biochemical or blood abnormalities commonly reported by individuals taking these treatments) and adherence to the allocated treatments among individuals receiving NFX or BZN for varying duration and dose, as compared with placebo
7. To explore differences in the impact of active treatments on the PCR among four subgroups of interest (geographical origin, T. cruzi discrete type unit found, parasitic load at baseline and age of participants).
8. To explore, among individuals treated with placebo, the level of agreement in the tests of parasitic load at baseline and during the follow up.

ELIGIBILITY:
Inclusion Criteria:

* Positive serology status to Trypanosoma cruzi
* No clinical signs of dilated cardiomyopathy

Exclusion Criteria:

* Unacceptable risk of re-infection, based on the investigators judgment
* Previous treatment with NFX or BZN
* History of peripheral neuropathy
* Health condition limiting the mobility, cognitive function or life expectancy within two years of the enrollment visit
* Pregnancy / Unwilling to use reliable contraceptive methods during childbearing age

Ages: 20 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 500 (Estimated)
Dates: Start 2015-08 (Actual); Primary Completion 2018-08 (Estimated); Study Completion 2019-02 (Estimated)

PRIMARY OUTCOMES:
Quantitative Polymerase Chain Reaction (qPCR) for Trypanosoma cruzi | 12 - 18 months after starting therapy
  Proportion of participants with at least one out of three positive tests (performed at least one week apart from each other)

SECONDARY OUTCOMES:
T. cruzi positive serology status | 12 months after starting therapy
  Proportion of participants with positive T. cruyzi serology status
Mean change in T. cruzi antibody titers | 12 months after starting therapy
  Mean change (before-after) in antibody readings as measured with ELISA serology

OTHER OUTCOMES:
Reported adverse reactions | 60 days after starting therapy
  Proportion of participants with at least one of the following a) Reporting hospitalization or inability to work b) Stopping study treatment because of adverse reactions /intolerance c) having abnormal levels of at least two biochemical or blood markers

CONTACTS AND LOCATIONS:
Overall Officials: Juan C Villar, MD, PhD, Principal Investigator — Universidad Autónoma de Bucaramanga
Locations (1):
- Fundación Oftalmológica de Santander - Clínica Ardila Lulle (FOSCAL), Bucaramanga, Santander Department, Colombia

REFERENCES:
- [Background] Villar JC, Perez JG, Cortes OL, Riarte A, Pepper M, Marin-Neto JA, Guyatt GH. Trypanocidal drugs for chronic asymptomatic Trypanosoma cruzi infection. Cochrane Database Syst Rev. 2014 May 27;2014(5):CD003463. doi: 10.1002/14651858.CD003463.pub2. PMID 24867876
- [Derived] Villar JC, Herrera VM, Perez Carreno JG, Vaquiro Herrera E, Castellanos Dominguez YZ, Vasquez SM, Cucunuba ZM, Prado NG, Hernandez Y. Nifurtimox versus benznidazole or placebo for asymptomatic Trypanosoma cruzi infection (Equivalence of Usual Interventions for Trypanosomiasis - EQUITY): study protocol for a randomised controlled trial. Trials. 2019 Jul 15;20(1):431. doi: 10.1186/s13063-019-3423-3. PMID 31307503